CLINICAL TRIAL: NCT02543879
Title: A Phase 1/1b Dose Escalation, Multicenter, Open-label, Safety, Pharmacokinetic and Pharmacodynamic Study of FT-1101 as a Single Agent and in Combination With Azacitidine in Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: Study of a Novel BET Inhibitor FT-1101 in Patients With Relapsed or Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1101-HEM-101
Record Dates: First submitted 2015-09-01; First posted 2015-09-07 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Non-Hodgkin Lymphoma
Keywords: AML; BET Inhibitor; FT-1101; Acute Leukemia; Myelodysplastic Syndrome; NHL; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Escalation FT-1101 (Experimental): Following a 3+3 dose escalation strategy, the first cohort of patients will be administered FT-1101 at 10 mg, oral capsules, once weekly on a continuous basis. Subsequent cohorts dose and frequency will be determined by investigators and sponsor following observations of previous cohorts. Dose escalation will continue until the MTD is determined.
  Interventions: Drug: FT-1101
- Dose Expansion FT-1101 (Experimental): Once the MTD is determined, the Recommended Phase 2 Dose (RP2D) will be identified. 3 Expansion cohorts of up to 20 patients each will be treated with the RP2D of FT-1101
  Interventions: Drug: FT-1101
- Dose Escalation FT-1101 + azacitidine (Experimental): Following a 3+3 dose escalation strategy, the first cohort of AML/MDS patients will be administered FT-1101 at approximately 50% or lower than the MTD identified for the single agent FT-1101. Subsequent cohorts dose will be determined by investigators and sponsor following observations of previous cohorts. Dose escalation will not exceed the dose determined to be the single agent MTD for that schedule.
  Interventions: Drug: FT-1101; Drug: Azacitidine
- Dose Expansion FT-1101 + azacitidine (Experimental): Once the MTD is determined, the Recommended Phase 2 Dose (RP2D) will be identified. 1 Expansion cohorts of up to 20 AML/MDS patients each will be treated with the RP2D of FT-1101 in combination with azacitidine.
  Interventions: Drug: FT-1101; Drug: Azacitidine

INTERVENTIONS:
Drug: FT-1101 — FT-1101 will be supplied as 5 mg, 20 mg or 100 mg capsules and will be administered per the protocol defined frequency and dose level
  Other Names: FT1101
Drug: Azacitidine — Azacitidine will be administered per site's standard of care
  Arms: Dose Escalation FT-1101 + azacitidine; Dose Expansion FT-1101 + azacitidine

SUMMARY:
This is an open-label, multicenter, dose-escalation Phase 1/1b study in patients with acute myelogenous leukemia (AML)/MDS or non-Hodgkin Lymphoma (NHL), intended to investigate safety, pharmacokinetics, and the pharmacodynamic effects of FT-1101 administered via one or more intermittent dosing schedules alone and in combination with azacitidine. Once the MTD has been established for a treatment cohort, up to 20 additional patients may be enrolled in up to 4 expansion cohorts each of select populations of patients with either AML/MDS or NHL at the recommended dose for future studies to confirm safety.

ELIGIBILITY:
Key Inclusion Criteria:

* Single agent (SA) Dose Escalation: Histologically or cytologically proven acute leukemia or high-risk MDS as defined by the World Health Organization (WHO) criteria and IPSS-R, respectively, that is relapsed or refractory (R/R) to standard therapy or for whom standard treatments are contraindicated, OR
* Mature B-Cell non-Hodgkin Lymphoma that is Relapsed/Refractory to standard therapy
* AML SA expansion group 1: histologically or cytologically proven AML with a FLT3 ITD or TKD mutation previously determined by local testing that is R/R to standard therapy or for whom standard treatments are contraindicated
* AML SA expansion group 2: histologically or cytologically proven AML with intermediate or unfavorable risk cytogenetics in the absence of a detectable FLT3 ITD or TKD mutation as previously determined by local testing that is R/R to standard therapy or for whom standard treatments are contraindicated
* NHL SA expansion: Mature B-cell NHL with the following histologies: primary mediastinal lymphoma, DLBCL, and B-cell lymphoma not specified that is R/R to standard therapy and for whom standard treatments are contraindicated or unavailable
* AML/MDS combination treatment (dose escalation and expansion): histologically or cytologically proven AML or MDS as defined by WHO criteria and IPSS-R, respectively, that is: R/R to standard therapy, or AML: who are unfit for, or unwilling to receive standard induction therapy, or MDS: eligible to receive azacitidine
* Patients ≥ 18 years old
* Good kidney and liver function
* No prior organ allograft
* For fertile men and women, agreement to use effective contraceptive methods duration of study participation and 90 days after

Key Exclusion Criteria:

* History of prior malignancy unless disease free for > or equal to 12 months or considered surgically cured.
* Patients with symptomatic central nervous system (CNS) metastases or other tumor location (such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture, etc.) necessitating an urgent therapeutic intervention, palliative care, surgery or radiation therapy
* Treatment with major surgery (requiring general anesthesia) within one month prior to study entry
* Previous treatment with any prior BET inhibitor therapy
* Patients unable to swallow oral medications, or patients with gastrointestinal conditions (e.g. malabsorption, gastric or small bowel resection, etc.) deemed to jeopardize intestinal absorption
* Congestive heart failure (New York Heart Association Class III or IV) or unstable angina pectoris. Previous history of myocardial infarction within 1 year prior to study entry, uncontrolled hypertension or uncontrolled arrhythmias
* Pulmonary disease (e.g. COPD, asthma, etc) that is not controlled (moderate to severe symptoms) with current medication
* Known HIV positivity
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within first 4 weeks of treatment
Dose Limiting Toxicities (DLT) | Within first 4 weeks of treatment
Recommended Phase 2 Dose (RP2D) | Participants to be followed for duration of participation, an expected average of 12 weeks

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | PK collected at multiple visits during the first 30 days of treatment
Peak Plasma Concentration (Cmax) | PK collected at multiple visits during the first 30 days of treatment
Time of peak plasma concentration (TMax) | PK collected at multiple visits during the first 30 days of treatment
Time for half of the drug to be absent in blood stream following dose (T 1/2) | PK collected at multiple visits during the first 30 days of treatment
Rate at which drug is removed from blood stream (CL/F) | PK collected at multiple visits during the first 30 days of treatment
Rate of drug distribution within the blood stream (Vd/F) | PK collected at multiple visits during the first 30 days of treatment
Observe patients for any evidence of anti-leukemic or anti-myelodysplastic activity of FT-1101 | Assessed for duration of participation, an expected average of 12 weeks

OTHER OUTCOMES:
Assessment of on-target activity of FT-1101, as determined by changes in PD biomarkers in bone marrow aspirates and/or peripheral blood | Assessed for duration of participation, an expected average of 12 weeks
To determine if there is any correlation between cancer-associated genetic alterations with response | Assessed for duration of participation, an expected average of 12 weeks
To evaluate PK/PD relationships in dose-escalation and dose-expansion cohorts | Assessed for duration of participation, an expected average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kelly, MD, Study Director — Forma Therapeutics, Inc.
Locations (8):
- United States (8):
  - Cedars Sinai, Los Angeles, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Levine Cancer Institute, Charlotte, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Crymes A, Evans MG, Jeyakumar D, Lou JJ, Zhao X, Rezk SA. Acute Myeloid Leukemia (AML) With T-Cell Differentiation Arising From Chronic Myelomonocytic Leukemia (CMML). Case Rep Hematol. 2024 Dec 14;2024:5584297. doi: 10.1155/crh/5584297. eCollection 2024. PMID 39734743